CLINICAL TRIAL: NCT02998112
Title: Fecal Microbiota Transplantation for Ulcerative Colitis Through Colonic Transendoscopic Enteral Tubing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Air Force Military Medical University, China (Other); First Hospital of Guangzhou (Unknown); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Zhongshan Hospital Xiamen University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMT-UC-121101
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Ulcerative Colitis
Keywords: fecal microbiota transplantation; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Placebo Comparator): 5-ASA 4g/day enema through TET for 1 week; 200ml saline infusion through TET for 3 times every other day in one week
  Interventions: Drug: Saline
- Study group (Experimental): 5-ASA 4g/day enema through TET for 1 week; 200ml fecal microbiota suspension infusion through TET for 3 times every other day in one week
  Interventions: Drug: fecal microbiota transplantation

INTERVENTIONS:
Drug: fecal microbiota transplantation — Fecal microbiota which was purified from fresh stool defecated by a healthy donor
  Arms: Study group
Drug: Saline
  Arms: control

SUMMARY:
To indicate the efficacy of Fecal microbiota transplantation (FMT) for the treatment of Ulcerative colitis (UC), The investigators design a multicenter, randomized controlled trial to perform FMT through colonic transendoscopic enteral tubing (TET) way, and evaluate the efficacy and safety of FMT for patients with moderate or severe UC.

DETAILED DESCRIPTION:
1. Patients with moderate to severe UC will be screened (Mayo>6）.
2. Participants will be divided into control and study groups by double blind.
3. Control group and study group will receive a colonic endoscopy evaluation. And a TET tube will be fixed at ileocecum.
4. Enema with 5-ASA 4g/day for 7days by TET will be performed as basic therapy for both control and study group. Study and control group will be given with fecal microbiota suspension and equal volume of saline by TET for three times every other day in one week.
5. The follow-up will be performed at 1 week, 4 weeks and 12 weeks after first treatment. All the participants will receive a endoscopy evaluation at 12 weeks. Clinical remission, clinical improvement and safety are the primary endpoint at 12 weeks; Intestinal microbiota changing is recognized as the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Active, moderate to severe severity (Mayo score more than 6)
* Safety using history of 5-ASA.
* Able to undergo endoscopy examination.

Exclusion Criteria:

* Immunosuppressive drugs and glucocorticoids using in 4 weeks
* Antibiotic using in 7 days
* High risk of toxic megacolon
* Colon cancer or neoplasia in pathophysiology
* Other severe diseases (eg: cardiovascular, respiratory, gastroenteral and kidney diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 12 weeks
  Total Mayo score less than 2 and no signal item more than 1
Clinical improvement | 12 weeks
  Total Mayo score decreased more than 3 or decreased more than 30%

SECONDARY OUTCOMES:
Intestinal microbiota changing | 12 weeks
  The change of intestinal microbiota composition after FMT compared with subject original microbiota and donor's microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929
- [Result] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Result] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Result] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986